CLINICAL TRIAL: NCT04504773
Title: Virtually Better: Using Immersive Virtual Reality to Treat Pediatric Anxiety
Brief Title: Using Immersive Virtual Reality to Treat Pediatric Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00210075
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-12

CONDITIONS: Specific Phobia; Specific Phobia, Situational; Specific Phobia, Animal; Specific Phobia, Natural Environment; Childhood Anxiety Disorder
Keywords: Exposure Therapy; Virtual Reality
MeSH Terms: conditions — Phobia, Specific | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Masking Description: Outcomes assessor is not involved in treatment, and will assess the severity of the participants anxiety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Exposure Therapy (Experimental): Participants will receive a single session of exposure therapy to address specific phobia that includes the use of virtual reality exposures.
  Interventions: Behavioral: Virtual Reality Exposure Therapy

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy — Participants will receive a single session of virtual reality exposure therapy that targets the participant's specific phobia stimuli.

SUMMARY:
Anxiety is a common and impairing problem for children. The principle treatment for pediatric anxiety involves facing a child's fears in a stepwise approach through a therapeutic exercise called exposures. While exposures are effective, some feared situations cannot be confronted in a clinician's office (e.g., heights, public speaking, storms). This poses a logistical challenge in treatment that: (1) takes time away from patient care, (2) leads clinicians to rely on imagined exposures, and/or (3) requires families to complete exposures outside of the therapy visits. This creates a burden for clinicians and families, and impedes treatment success. Immersive virtual reality (VR) presents an innovative solution that allows children to face fears without leaving the clinician's office. While VR has been used to distract children during painful medical procedures, it has not been well examined as a primary treatment for pediatric anxiety. This study proposes to examine the effectiveness and acceptability of using immersive VR exposures to treat children and adolescents with specific phobias.

ELIGIBILITY:
Inclusion Criteria:

* 8-17 years (inclusive),
* meet diagnostic criteria for one or more phobias on a structured diagnostic interview (ADIS-C/P). This specifically includes natural environments (e.g., storms, heights) and/or situational settings (e.g., airplanes, public speaking).
* be fluent in English.

Exclusion Criteria:

* unable to complete rating scales, or
* attend study visits.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Clinical Severity Rating (CSR) of Targeted Specific Phobia on Anxiety Disorder Interview Schedule for Children and Parents (ADIS-C/P) | 1 week after virtual reality exposure therapy session
  The ADIS-C/P CSR for the Specific Phobia is a single item rating that is made by a clinician. Scores are made on a 9-point scale that ranges from 0 (Not at all) to 8 (Very, very much). A score of 4 or greater considered to be indicative of a psychiatric disorder.

SECONDARY OUTCOMES:
Screen for Childhood Anxiety and Related Disorders-Parent Report (SCARED-P) | 1 week after virtual reality exposure therapy session
  Parent-reported rating of child anxiety that consists of 41-items. Items are rated on a 3-point scale that ranges from 0 (Not True) to 2 (Very True). The total score ranges from 0 to 82, with a total score of 25 or greater may indicate the presence of an anxiety disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F. McGuire, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No